CLINICAL TRIAL: NCT06761144
Title: Pulmonary Thromboembolism in Cancer Patients: Early Rule-out From the Emergency Department
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PS-23-01; RC-2022-2773366 (Other Grant/Funding Number: Ricerca Corrente 2022-2024 - Italian Ministry of Health)
Record Dates: First submitted 2024-12-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Thromboembolisms
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulmonary thromboembolism is a frequent complication of cancer; in some cases, it is diagnosed occasionally during diagnostic examinations as part of the regular follow-up of the disease. Not all patients diagnosed with thromboembolism present symptoms; therefore, after appropriate investigations during observation in the emergency room and/or a short hospitalisation in Emergency Medicine, they could be discharged home, avoiding lengthy hospitalisations that would have a considerable impact on their health and psychological condition.

The goal of this observational study is to compare the efficacy of several assessment scales for use by physicians to identify patients at low risk of developing serious complications of pulmonary embolism within 30 days of diagnosis, in order to be able to identify a group of low-risk patients who could be discharged early from the emergency department/emergency medicine safely.

What does participation in this study entail compared to the normal care you receive and what are your responsibilities as a participant? At the time of patient enrolment in the emergency room/emergency medicine, the data necessary for the calculation of 6 scoring systems will be collected, which will take approximately 5 minutes.

The patient enrolled in the study will be contacted by telephone in order to assess the state of health; the call will take approximately 1 minute and will take place 30 days after access to the emergency room.

Participation in the study does not entail any obligation or restriction, nor will it be charged for.

DETAILED DESCRIPTION:
Cancer patients are at increased risk of developing thromboembolic complications, including pulmonary thromboembolism (PTE), with an annual incidence of 1:200. Not all patients with PTE present with symptoms suggestive of the disease, and nowadays, thanks in part to the technological development of radiological techniques that make it possible to visualise as far as the subsegmental branches of the pulmonary vasculature, the diagnosis of pulmonary embolism is steadily increasing. Therefore, we are increasingly seeing the diagnosis of Incidental Pulmonary Embolism (IPE), defined as 'an unsuspected pulmonary artery filling defect identified during CT scans performed for other reasons, usually during screening and follow-up of cancer pathology'. Patients with IPE are often asymptomatic, although in some cases, further investigation of the history and complaints reported by the patient may reveal some symptoms compatible with PTE.

The incidence of IPE in cancer patients ranges from 1.6 to 7.3%. In this study, patients who presented to the Emergency Department during the period from 01.01.2015 to 31.12.2019 will be consecutively enrolled in a retrospective manner and prospectively patients presenting to the Emergency Department for a period of two years from the approval of the study by the Ethics Committee and subsequent clearance by the Director General with a diagnosis of PTE in the course of active onco-haematological disease (pathology followed in an oncological/haematological and/or metastatic setting).

A 30 day follow-up will be carried out in order to record any major adverse events, like death, respiratory failure, or re-hospitalisation.

The study is observational, non-interventional. Patients will be treated according to clinical practice in accordance with the judgement of the physician.

The primary objective is to evaluate existing and used prognostic scores (HESTIA, PESI, sPESI, POMPE-C, EPIPHANY Index, RIETE) in oncological patients with incidental pulmonary embolism in order to identify the one with the greatest effectiveness in identifying patients at low risk of major adverse events at 30 days, and therefore safely discharged early from the emergency department.

The secondary objective is to identify, in the group of cancer patients with pulmonary embolism (incidental and symptomatic), which score among those used has the best performance in identifying patients at low risk of major adverse events at 30 days, in order to identify a group of patients who can be discharged early and safely.

The outcome to be assessed is 30-day mortality in patients identified as low risk with the scores used. In addition, evaluate a composite endpoint at 30 days: hospitalisation for PTE diagnosis-related problems/respiratory failure-related illness/mortality at 30 days.

It should be noted that the diagnosis of acute respiratory failure will be made according to the diagnostic criteria known in the literature. This diagnosis imposes the need for oxygen therapy, so the patient with respiratory failure will not be discharged home, necessarily requiring hospitalisation, which is an adverse event for the proposed study.

Outcomes will be assessed using computerised records and PS reports. Patients over 18 years of age attending the General Hospital / Emergency Medicine IRCCS AOU of Bologna Policlinico di S.Orsola with a diagnosis of PTE and onco-haematological pathology will be included. The duration of the study is estimated to be 3 years: 6 months for retrospective data collection, 24 months for prospective enrolment and 6 months for data processing.

It should be noted that patients will be enrolled at the first admission to the Emergency Department, therefore they will be in charge of the Emergency Department and not in an in-patient setting. The enrolled patients could be retained in the OBI regime (always afferent to the Emergency Department) to complete the basic diagnostic-therapeutic procedure before eventual admission to a medical, intensive-sub-intensive ward or discharge to home. Any admission to Emergency Medicine, following discharge from the Emergency Department, will be considered as admission to an internist environment.

Patient characteristics will be reported as mean +/- standard deviation for continuous variables and as numerosity and frequency for categorical variables. Sensitivity, specificity, positive and negative predictive values will be calculated for each score. Monovariate statistics using Kaplan Meier curves will be used to assess the association of each score with 30-day mortality. In addition, ROC (Receiver-operating Characteristic) curve analysis will be used to evaluate the performance of each score. Statistical significance will be defined for values of p<0.05 and analyses will be conducted using SPSS version 28 software (IBM Corp., Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of pulmonary embolism (symptomatic and/or incidental)
* Active onco-haematological disease (disease followed in oncological/haematological and/or metastatic setting)
* Informed consent to the study

Exclusion Criteria:

* Patients returning to the Emergency Department for complications related to previously diagnosed pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active oncohematological pathology, over 18 years of age, with a diagnosis of pulmonary embolism attending the Emergency Department of the IRCSS Azienda Ospedaliero-Universitaria di Bologna
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07-13 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate mortality in patients at low risk of major adverse events (death/respiratory failure/hospitalisation) | From enrollment to the follow-up at 30 days
  The primary objective is to evaluate the already existing and used prognostic scores (HESTIA, PESI, sPESI, POMPE-C, EPIPHANY Index, RIETE) in cancer patients with incidental pulmonary embolism in order to identify the one with the greatest effectiveness for identifying patients at low risk of major adverse events at 30 days, who can therefore be discharged early and safely from the emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Tubertini, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- Eleonora Tubertini, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No